CLINICAL TRIAL: NCT06615895
Title: The Effectiveness of Telehealth-Based Family-Centered Early Intervention: Enhancing Sensory Inputs Activities on Vision and Posture-Movement Performance
Brief Title: The Effectiveness of Telehealth-Based Family-Centered Early Intervention
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMU-JIRB N202407062; 113HCP-04 (Other Grant/Funding Number: Shuang Ho Hospital)
Record Dates: First submitted 2024-09-22; First posted 2024-09-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2024-09

CONDITIONS: Children Receiving Early Intervention; Visual Perception Performance; Effects of Posture and Movement
Keywords: sensory processing disorders; Telehealth-health; Family-Centered

STUDY DESIGN:
Intervention Model Description: Subjects are assigned to the "telehealth group" or the "waiting group".
  The "telehealth group" participates in an online video course for 6 weeks. The therapist will provide online video courses 3-5 times a week and record the implementation on the online platform every week. The course includes action plans, two Lateral integration/cross-midline, vestibular system, visual perception, opto-motor integration, eye movements, core strength activities and balance ability, etc.
  The "waiting group" is to provide explanation of course objectives and wait for 6 weeks after explaining the objectives of this research in the first course.
Who Masked: Outcomes Assessor
Masking Description: Assessment tests are conducted before and after the intervention. The assessor is the same person, who is a single-blind and professionally trained therapist who does not know the group assignment of the case.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Telehealth group (Experimental): An online video course for 6 weeks. The therapist will provide online video courses 3-5 times a week and record the implementation on the online platform every week. The course includes action plans, two Lateral integration/cross-midline, vestibular system, visual perception, opto-motor integration, eye movements, core strength activities and balance ability, etc.
  Interventions: Behavioral: Telehealth home activity
- Waiting group (No Intervention): The "waiting group" was provided with an explanation of the objectives of the course. After the objectives of the study were explained in the first course, they waited for 6 weeks before receiving remote intervention.

INTERVENTIONS:
Behavioral: Telehealth home activity — Several course activities with diverse sensory modalities are provided a week. Caregivers or caretakers need to help children participate in the course content and implement relevant suggestions at least 3-5 times a week for six weeks. The research will be conducted on an online platform. Course announcements, reminders and confirmation of work execution, through caregivers' feedback records, urge caregivers to engage in parent-child games related to sensory integration and integrated into life at home. Such high-frequency, short-term sensory activities will be adapted to the equipment available at home. It will mainly focus on movement planning, bilateral integration/crossing the midline, vestibular system , visual perception, visual-motor integration, eye movements, core strength activities and Activities focused on balance ability.
  Arms: Telehealth group

SUMMARY:
Background: Children with developmental delays or sensory processing disorders (SPD) face challenges in processing and integrating sensory information from their environment, which can lead to behavioral, learning, and social issues. Visual-vestibular stimulation activities target fundamental abilities such as balance, coordination, and sensory processing, which are crucial for many developmental areas. Past literature supports the use of digital media as a medium to provide ongoing home-based occupational therapy interventions for children who are unable to receive in-person treatment, with opportunities for caregiver-guided interventions. Therefore, this project is designed based on the "1001 Children's Therapy Activities" model as the foundation for behavioral intervention, combining parent and child participation in play to establish effective home activities and execution, aiming to enhance children's visual perception and posture-movement performance, thereby improving learning outcomes.

Objective: To investigate the impact of a "Telehealth Visual and Vestibular Home Program" that integrates parent and child activity participation on children's visual perceptual performance and posture-movement effects.

Method: Caregivers of children attending early intervention clinics at a teaching hospital in northern Taiwan are recruited and randomly assigned to either a remote group (N=30) or a waitlist group (N=30). The remote group receives a 6-week visual and vestibular home course; the waitlist group will participate after a 6-week. Assessments using the Developmental Test of Visual Perception (DTVP-2), the Movement Assessment Battery for Children, Second Edition (MABC-2), and a course satisfaction questionnaire are conducted before and after the intervention.

Data Analysis: Basic data are presented using descriptive statistics, and t tests are used to compare pre- and post-training assessment mean values. Statistical analysis is performed using SPSS 26.0, with a significance level set at Alpha<0.05.

DETAILED DESCRIPTION:
Past literature supports that digital media can be used as a medium to provide continuous interventional home-based occupational therapy for children who cannot receive physical therapy, and has the opportunity to guide the intervention through caregivers (Marino et al., 2020), using different visual and vestibular senses. For intervention factors, a home-based teaching model is designed to meet the needs of high-frequency supervision and feedback established by habits. It can respond appropriately and immediately to difficulties and adjust settings. In addition to providing timely assistance, individual consultations can also be provided on the online platform. , based on the capabilities of individual families or caregivers, as well as the child's own temperament and abilities, we provide exclusive technical advice to minimize difficulties and make the use of strategies more successful to help establish good home activities. Through the remote home teaching model, children's execution can be increased, including action planning, bilateral coordination, vestibular processing, visual perception, visual-motor integration and eye movement, thereby increasing the improvement of children's visual perception, posture and movement ( Božanić Urbančič et al., 2023; Wiener-Vacher et al., 2013; Yılmaz & Önal, 2021). For children who receive early treatment, caregivers often fail to provide ideal guidance despite intentional guidance. They are unable to provide appropriate home therapy activities according to the children's abilities and needs, and they also deviate from the games that children should participate in during their development. Therefore, through professional and standardized intervention models, subtle changes and learning in daily life are established in this way, promoting the quality of their visual movements and increasing learning performance.

In the clinical practice of early childhood education in our hospital, there is a lack of home treatment programs for early childhood education. This study intends to use the specific model of "1001 Children's Treatment Activities" as the basis for intervention in behavior change, combined with the participation of parents and children in games, to establish the basis for children's effective treatment. Good home activities and execution can improve children's visual perception, posture and movements, thereby improving learning performance.

ELIGIBILITY:
Inclusion Criteria:

* (1) Children currently receiving early treatment; (2) Children with caregivers who need to establish a home treatment plan; (3) Children who can cooperate with the trial process and complete homework at home, and have completed at least 5/6 of the training; (4) There is an Internet connection;

Exclusion Criteria:

* (1) Children's medical records show a diagnosis of central nervous system injury (such as cerebral palsy, brain trauma, epilepsy, cortical blindness), rare disease diagnosis (such as William's disease, Down syndrome); (2) Children under 3 years old , 7 years old and above; (3) The caregiver cannot communicate in Chinese.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Children's sensory integration function assessment scale (preschool version) | before and after the intervention, study completion, an average of 6 weeks
  In order to diagnose children with abnormal sensory integration in Taiwan, it covers seven dimensions of disorders and the phenomenon of sensory unintegration, with a total of 98 questions: posture and movement, integrated movement sequence on both sides, sensory discrimination, sensory adjustment, sensory search, and attention. and activity level, emotional/behavioral reactions, using a five-point scale. The higher the score, the worse the sensory integration, that is, the more obvious the disorder characteristics are. The test-retest reliability of each subscale is between .82 and .94; internal Consistency reliability ranges from .80 to .94

SECONDARY OUTCOMES:
Developmental Test of Visual Perception (DTVP-2) | before and after the intervention, study completion, an average of 6 weeks
  A paper-and-pencil test that assesses the visual perception and visual movement integration abilities of children aged 4 to 12 years and 11 months, including hand-eye coordination, spatial position, imitation, subject-background distinction, spatial relationship, visual gestalt, optomotor speed, and shape constancy. Internal consistency>0.7, reliability and validity 0.78-0.91
Movement Assessment Battery for Children for Children, Second Edition ( MABC-2) | before and after the intervention, study completion, an average of 6 weeks
  The age of the test is 3-16 years and 11 months. It evaluates the ability of hand dexterity, aiming and receiving objects, and balance. It uses the upper limb movement coordination subtest. It has good reliability and validity, and internal consistency (Internal consistency) α =0.90, test-retest reliability (Test-retest reliability) is ICC= 0.97, minimal detectable change (MDC) is 0.28 points, and minimal important difference (MID) is 2.36 to 2.50
the number of adverse reactions and side effects | After the intervention, study completion, an average of 6 weeks
  After the intervention, ask whether there are any adverse reactions or side effects, such as aches, pains, injuries, etc., and record the number of occurrences in the case record form
Course satisfaction questionnaire | After the intervention, study completion, an average of 6 weeks
  A self-made questionnaire based on the course content has a total of 12 questions, using a 5-point scale to collect data on caregivers' acceptance of the course, implementation effectiveness, and feedback on course implementation and changes in children.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University Shuang Ho Hospital, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wiener-Vacher SR, Hamilton DA, Wiener SI. Vestibular activity and cognitive development in children: perspectives. Front Integr Neurosci. 2013 Dec 11;7:92. doi: 10.3389/fnint.2013.00092. eCollection 2013. PMID 24376403
- [Background] Schoen SA, Lane SJ, Mailloux Z, May-Benson T, Parham LD, Smith Roley S, Schaaf RC. A systematic review of ayres sensory integration intervention for children with autism. Autism Res. 2019 Jan;12(1):6-19. doi: 10.1002/aur.2046. Epub 2018 Dec 12. PMID 30548827
- [Background] Önal, G., Güney, G., Gün, F., & Huri, M. (2021). Telehealth in paediatric occupational therapy: a scoping review. International Journal of Therapy and Rehabilitation, 28(7), 1-16.
- [Background] Moghadam, S. F., Haghgoo, H. A., Pishyareh, E., Bakhshi, E., Rezazadeh, N., Rostami, R., & Sadeghi, V. (2018). Vestibular therapy improved motor planning, attention, and balance in children with attention deficit hyperactivity disorders: a randomized controlled trial. Phys Med Rehabil Res, 3(2), 1-6.
- [Background] Mikami M, Hirota T, Takahashi M, Adachi M, Saito M, Koeda S, Yoshida K, Sakamoto Y, Kato S, Nakamura K, Yamada J. Atypical Sensory Processing Profiles and Their Associations With Motor Problems In Preschoolers With Developmental Coordination Disorder. Child Psychiatry Hum Dev. 2021 Apr;52(2):311-320. doi: 10.1007/s10578-020-01013-5. PMID 32529540
- [Background] Marino F, Chila P, Failla C, Crimi I, Minutoli R, Puglisi A, Arnao AA, Tartarisco G, Ruta L, Vagni D, Pioggia G. Tele-Assisted Behavioral Intervention for Families with Children with Autism Spectrum Disorders: A Randomized Control Trial. Brain Sci. 2020 Sep 18;10(9):649. doi: 10.3390/brainsci10090649. PMID 32961875
- [Background] Hung Kn G, Fong KN. Effects of telerehabilitation in occupational therapy practice: A systematic review. Hong Kong J Occup Ther. 2019 Jun;32(1):3-21. doi: 10.1177/1569186119849119. Epub 2019 May 27. PMID 31217758
- [Background] Huang CY, Huang TY, Koh CL, Yu YT, Chen KL. The Movement Assessment Battery for Children Second Edition in Ages 3 to 6 Years: A Cross-Cultural Comparison for Children in Taiwan. Phys Ther. 2024 Jan 1;104(1):pzad146. doi: 10.1093/ptj/pzad146. PMID 37883453
- [Background] Blanche, E. I., Giuffrida, C., Hallway, M., Edwards, B., & Test, L. A. (2021). An Evidence-based Guide to Combining Interventions with Sensory Integration in Pediatric Practice. Routledge.